CLINICAL TRIAL: NCT03751631
Title: A Double-Masked, Active-Controlled Study of the Safety and Efficacy of Phenylephrine 2.5%-Tropicamide 1% Ophthalmic Solution Administered With a Microdose Dispenser for Dilation of the Pupil
Brief Title: Safety and Efficacy of Phenylephrine 2.5%-Tropicamide 1% Microdose Ophthalmic Solution for Pupil Dilation
Acronym: MIST-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: EYN-MYD-TP-31
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-01

CONDITIONS: Mydriasis
MeSH Terms: conditions — Mydriasis | interventions — Tropicamide; Phenylephrine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This trial was a double-masked, active-controlled, cross-over superiority study evaluating the efficacy of the fixed combination drug vs. the drug's 2 individual components. All participants in the trial were to receive each of the 3 drugs.
Who Masked: Participant, Outcomes Assessor
Masking Description: There were no differences in the presentation of drug administered and all study personnel conducting ophthalmic assessments after drug administration were masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1-TR/PE, 2-TR, 3-PE (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)
- 1-TR/PE, 2-PE, 3-TR (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)
- 1-TR, 2-TR/PE, 3-PE (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)
- 1-TR, 2-PE, 3-TR/PE (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)
- 1-PE, 2-TR/PE, 3-TR (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)
- 1-PE, 2-TR, 3-TR/PE (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the study drug in each eye.
  Interventions: Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE); Drug: Tropicamide 1% ophthalmic solution (TR); Drug: Phenylephrine 2.5% ophthalmic solution (PE)

INTERVENTIONS:
Drug: Tropicamide 1%-Phenylephrine 2.5% ophthalmic solution (TR/PE) — Fixed combination tropicamide 1%-phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser
  Other Names: Mydcombi
Drug: Tropicamide 1% ophthalmic solution (TR) — Tropicamide 1% ophthalmic solution administered with the Optejet microdose dispenser
Drug: Phenylephrine 2.5% ophthalmic solution (PE) — Phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser

SUMMARY:
This study evaluated pupil dilation after administration of fixed combination tropicamide-phenylephrine (TR/PE) vs. phenylephrine (PE) alone and tropicamide (TR) alone. Participants attended 3 visits. At each visit, after baseline measurements, 1 of the 3 drugs was administered to both eyes, then pupil dilation and safety assessments were performed at specific time intervals.

DETAILED DESCRIPTION:
Volunteer participants were screened for study eligibility during a Screening Visit and enrolled after signing the study-specific informed consent form. Subjects meeting all inclusion/exclusion criteria were scheduled for 3 treatment visits, which were at least 2 days, but no more than 7 days apart. At each treatment visit, baseline measurements were taken, then 1 of the 3 study drugs was administered to both eyes (each participant's drug administration sequence was randomly determined). Afterwards, efficacy and safety assessments were performed at 20, 35, 50, 65, 80, 120, and 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent and return for all study visits
* Photopic pupil diameter <= 3.5 mm in each eye

Exclusion Criteria:

* Allergy to phenylephrine hydrochloride, tropicamide, or benzalkonium chloride
* History of benign prostatic hyperplasia
* Use of a benzodiazepine, monoamine oxidase inhibitor, tricyclic antidepressant, anticonvulsant, or cholinergic drug
* History of closed-angle glaucoma
* Anatomically narrow anterior chamber angles
* Ocular surgery or laser treatment of any kind
* History of chronic or acute uveitis
* History of traumatic iritis or hyphema
* History of traumatic mydriasis or angle recession
* History of heterochromia
* Irregularly-shaped pupil secondary to ocular trauma or congenital defect.
* History of neurogenic pupil disorder
* History of anterior chamber intraocular lens (IOL) or iris-fixated IOL
* History of iris surgery, iris atrophy, or iris-cornea apposition/touch
* Unwilling or unable to discontinue use of contact lenses at treatment visits.
* Current active eye disease for which topical or systemic ophthalmic medication is necessary, except for dry eye disease managed using artificial tears.
* Presence of a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment and/or follow-up
* Pregnancy or lactation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho Ianchulev, MD, MPH, Study Director — Eyenovia Inc.
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 patients signed the study informed consent form and were screened for eligibility between October 31, 2018 and November 16, 2018 at a clinical research center located in Cypress, California.
Pre-assignment Details: 64 of the 70 participants enrolled initiated treatment. Of those who did not initiate treatment, 4 failed to meet all study eligibility criteria, 1 was exited during screening due to behavioral issues, and 1 was exited after screening (before treatment) because the investigator believed the required number of subjects had initiated treatment.
Units Other Than Participants: eyes
Groups:
- TR/PE - TR - PE: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Tropicamide 1%-Phenylephrine 2.5%; 2nd Treatment Day - Tropicamide 1%; 3rd Treatment Day - Phenylephrine 2.5%. Each drug was administered with the Optejet microdose dispenser.
- TR/PE - PE - TR: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Tropicamide 1%-Phenylephrine 2.5%; 2nd Treatment Day - Phenylephrine 2.5%; 3rd Treatment Day - Tropicamide 1%. Each drug was administered with the Optejet microdose dispenser.
- TR - TR/PE - PE: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Tropicamide 1%; 2nd Treatment Day - Tropicamide 1%-Phenylephrine 2.5%; 3rd Treatment Day - Phenylephrine 2.5%. Each drug was administered with the Optejet microdose dispenser.
- TR - PE - TR/PE: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Tropicamide 1%; 2nd Treatment Day - Phenylephrine 2.5%; 3rd Treatment Day - Tropicamide 1%-Phenylephrine 2.5%. Each drug was administered with the Optejet microdose dispenser.
- PE - TR/PE - TR: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Phenylephrine 2.5%; 2nd Treatment Day - Tropicamide 1%-Phenylephrine 2.5%; 3rd Treatment Day - Tropicamide 1%. Each drug was administered with the Optejet microdose dispenser.
- PE - TR - TR/PE: Participants were administered the assigned study drug in each eye on separate days in the following order: 1st Treatment Day - Phenylephrine 2.5%; 2nd Treatment Day - Tropicamide 1%; 3rd Treatment Day - Tropicamide 1%-Phenylephrine 2.5%. Each drug was administered with the Optejet microdose dispenser.
Period: Overall Study
Arm/Group | TR/PE - TR - PE | TR/PE - PE - TR | TR - TR/PE - PE | TR - PE - TR/PE | PE - TR/PE - TR | PE - TR - TR/PE
Started | 10; 20 eyes | 11; 22 eyes | 11; 22 eyes | 11; 22 eyes | 10; 20 eyes | 11; 22 eyes
Received 1st Drug in Sequence | 10; 20 eyes | 11; 22 eyes | 11; 22 eyes | 11; 22 eyes | 10; 20 eyes | 11; 22 eyes
Received 2nd Drug in Sequence | 10; 20 eyes | 11; 22 eyes | 10; 20 eyes | 10; 20 eyes | 10; 20 eyes | 11; 22 eyes
Received 3rd Drug in Sequence | 10; 20 eyes | 11; 22 eyes | 10; 20 eyes | 10; 20 eyes | 10; 20 eyes | 11; 22 eyes
Completed | 10; 20 eyes | 11; 22 eyes | 10; 20 eyes | 10; 20 eyes | 10; 20 eyes | 11; 22 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 1; 2 eyes | 1; 2 eyes | 0; 0 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were administered each of the 3 assigned drugs on 3 separate days in the clinic (drug administration sequence was equally randomized across 6 possible administration sequences).
Arm/Group | All Participants
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 35
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 64
Iris color category [Count of Participants; unit: Participants] — Dark = Brown/black irides Light = All other colors
  Participants
    Dark | 54
    Light | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Pupil Diameter From Baseline
Description: Difference in 35-minute pupil diameter vs. baseline measured using pupillometry in highly photopic conditions.
  Pupil diameter is reported in millimeters. For the change in pupil diameter, larger measurements indicate a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- TR/PE - Right Eye: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered to the right eye with the Optejet microdose dispenser
- TR/PE - Left Eye: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered to the left eye with the Optejet microdose dispenser
- TR - Right Eye: Tropicamide 1% ophthalmic solution administered to the right eye with the Optejet microdose dispenser
- TR - Left Eye: Tropicamide 1% ophthalmic solution administered to the left eye with the Optejet microdose dispenser
- PE - Right Eye: Phenylephrine 2.5% ophthalmic solution administered to the right eye with the Optejet microdose dispenser
- PE - Left Eye: Phenylephrine 2.5% ophthalmic solution administered to the left eye with the Optejet microdose dispenser
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | TR - Right Eye | TR - Left Eye | PE - Right Eye | PE - Left Eye
Number analyzed (Participants) | 62 | 62 | 62 | 62 | 62 | 62
millimeters
  Baseline pupil diameter | 2.672 (0.5673) | 2.583 (0.4674) | 2.657 (0.6016) | 2.569 (0.5211) | 2.651 (0.5749) | 2.584 (0.5344)
  35-minute pupil diameter | 7.301 (0.8943) | 7.329 (0.9771) | 6.762 (0.8619) | 6.690 (0.8682) | 3.388 (0.8950) | 3.552 (0.9340)
  Change in 35-minute pupil diameter | 4.629 (0.8343) | 4.746 (0.8173) | 4.105 (0.7207) | 4.121 (0.6839) | 0.737 (0.7939) | 0.969 (0.8943)

2. Other Pre Specified Outcome: Percentage of Eyes Achieving Pupil Diameter 6.0 mm or Larger After Receipt of Each Medication
Description: The percent of eyes with pupil diameter 6.0 mm or larger as measured using pupillometry in highly photopic conditions. As this is a cross-over study, each of the 62 participants received each medication. Data is reported separately for the right and left eyes of the 62 participants. A higher percentage indicates a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | TR - Right Eye | TR - Left Eye | PE - Right Eye | PE - Left Eye
Number analyzed (Participants) | 62 | 62 | 62 | 62 | 62 | 62
Number analyzed (Eyes) | 62 | 62 | 62 | 62 | 62 | 62
percentage of eyes | 95.2 | 93.5 | 79.0 | 77.4 | 1.6 | 1.6

3. Other Pre Specified Outcome: Percentage of Eyes Achieving Pupil Diameter 7.0 mm or Larger After Receipt of Each Medication
Description: The percent of eyes with pupil diameter 7.0 mm or larger as measured using pupillometry in highly photopic conditions. As this is a cross-over study, each of the 62 participants received each medication. Data is reported separately for the right and left eyes of the 62 participants. A higher percentage indicates a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | TR - Right Eye | TR - Left Eye | PE - Right Eye | PE - Left Eye
Number analyzed (Participants) | 62 | 62 | 62 | 62 | 62 | 62
Number analyzed (Eyes) | 62 | 62 | 62 | 62 | 62 | 62
percentage of eyes | 67.7 | 67.7 | 43.5 | 41.9 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over each subject's study participation period, which was a maximum of 14 days
Groups:
- Tropicamide/Phenylephrine: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser
- Tropicamide: Tropicamide 1% ophthalmic solution administered with the Optejet microdose dispenser
- Phenylephrine: Phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser
Arm/Group | Tropicamide/Phenylephrine | Tropicamide | Phenylephrine
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64 | 0/62
Other Adverse Events (participants affected / at risk) | 2/62 | 4/64 | 4/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tropicamide/Phenylephrine (N=62) | Tropicamide (N=64) | Phenylephrine (N=62)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT03751631/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03751631/SAP_001.pdf
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT03751631/ICF_002.pdf